CLINICAL TRIAL: NCT02897024
Title: A Comparison: High Intense Periodic vs. Every Week Therapy in Children With Cerebral Palsy (ACHIEVE)
Acronym: ACHIEVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Jill Heathcock, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016N0031
Record Dates: First submitted 2016-09-07; First posted 2016-09-12 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Motor Impairments
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual weekly (Active Comparator): Usual weekly physical therapy is 1 hours of therapy one day per week for 40 weeks.
  Interventions: Other: Physical Therapy
- High intensity periodic (Experimental): High intensity periodic physical therapy is 2 hours of therapy 5 days a week for 2 weeks, followed by an 18 week break, followed by another bout of high intensity therapy for 2 hours of therapy every weekday for two 10-consecutive-weekdays, followed by another 18 week break from therapy.
  Interventions: Other: Physical Therapy

INTERVENTIONS:
Other: Physical Therapy — One-on-one physical therapy sessions (one therapist and one patient). Principles of motor learning used include repetition, task-specificity, active practice, generalization of skills, errors, structured practice, and developmentally appropriate feedback with sufficient time to practice.

SUMMARY:
The ACHIEVE study is a comparison of the effectiveness of 2 intensities of physical therapy treatment for children with Cerebral Palsy in an outpatient physical therapy setting. High intensity periodic is 2 hours of focused and high intense treatment per weekday for 4 weeks. In comparison, usual weekly is considered standard of care; although both dosing models are used clinically for children with CP. Participants are assign to the treatment group at random. Participant who are unable to consent to randomization are allowed to chose a treatment group.

DETAILED DESCRIPTION:
The overall goal of this project is to compare the effectiveness of high intense periodic and usual weekly therapy in treating Cerebral Palsy (CP) in children 2-8 years of age for motor rehabilitation. In this prospective randomized controlled trial (RCT), 108 children ages 2 to 8 years of age with CP will be enrolled and assigned to one of 2 service delivery models: 1 hour per day, 1 x per week for 40 weeks (usual weekly); and 2 hours every weekday for two 10-consecutive-weekdays (total 4 weeks), for a repeated "periodic" bout (high intense periodic). Participants unable to consent to randomization are allowed to chose a treatment group. All patients enrolled in ACHIEVE will also have 1 hour per month of Physical Therapy Consultation (PTC) during the treatment period of 40 weeks (9 months). PTCs provide monthly motor skill monitoring, consultation, and home therapy program progression. Outcome evaluations will be performed by blinded evaluators at baseline (month 0, before treatment), month 9 for all patients to assess short term effects, and at months 12 and 18 for patients to assess long term effects. Parent surveys will be collected at 0, 4.5, and 9 months only (PC-2). Short-term and long-term effects will be analyzed to determine individual differences in children's response to intensity. A subset will be analyzed at 12 and 18 month.

ELIGIBILITY:
Inclusion Criteria:

* 2 to 8 years of age at initiation of treatment
* a diagnosis of motor delay or CP in GMFCS levels 1-V
* ability to tolerate a 2 hour therapy session based on parent report and evaluating therapists.

Exclusion Criteria:

* uncontrollable seizures or any co-morbid condition that prevents full participation during treatment sessions
* participation in another daily treatment program in the last 6 months
* auditory or visual conditions that prevent full participation during treatment sessions
* Progressive neurological disorder with no potential for improvement.
* Recent surgery where physical therapy is contraindicated.

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Change in Gross Motor Function Measure (GMFM)-88 | Baseline (pre-treatment) and 9 months 12 months, and 18 months following initiation of treatment.
  GMFM evaluates change in gross motor function over time or with intervention in children

SECONDARY OUTCOMES:
Change in Goal Attainment Scaling (GAS) | Baseline (pre-treatment) and 9 months 12 months, and 18 months following initiation of treatment.
  GAS creates patient, family, and clinical anchors as the external criterion for improvement by establishing activity or participation goals that reflect what an individual, family, and clinician consider meaningful or relevant.The GAS method allows for goals to be defined at different levels of mastery and assigned numerical values for score calculation, similar to a Likert scale. The scale will have 5 points representing different levels of mastery of the individual patient's goal. A score of -2 represents baseline, -1 less change than expected, 0 for the expected level of change, and +1 and +2 for achievement of more change than expected. To attempt to ensure ordinality, each level on the scale will be described and will reflect a single dimension of change that is measureable, achievable, and relevant
Change in Bayley Scales of Infant Development III | Baseline (pre-treatment) and 9 months 12 months, and 18 months following initiation of treatment.
  The Bayley Scales of Infant and Toddler Development-Third Edition is an individually administered test designed to assess developmental functioning of infants and toddlers. The Bayley-III assesses development in five areas: cognitive, language, motor, social-emotional, and adaptive behavior.
Change in Pediatric Evaluation and Disability Inventory (PEDI) | Baseline (pre-treatment) and 9 months 12 months, and 18 months following initiation of treatment.
  Administered as a parent survey. The PEDI is a descriptive measure of a child's current functional performance and can track changes over time. The PEDI measures both capability and performance of functional activities in three content domains: self-care, mobility, and social function.It can be used as a comprehensive clinical assessment of key functional capabilities and performance in children between the ages of six months and seven years.

OTHER OUTCOMES:
Change in Pediatric Outcomes Questionnaire (PODCI) | Collected at 0, 4.5 and 9 months (during the treatment period)
  Parent survey to assess patients under the age of 19 years for overall health, pain, and ability to participate in normal daily activities, as well as more vigorous activities typically associated with young people. The target populations are children and adolescents ages 2-18 years with general health problems, specifically any problems related to bone and muscle conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Heathcock, MPT, PhD, Principal Investigator — Ohio State University
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Maus E, Sansuchat LA, Tripathi T, Heathcock JC. Mostly Mothers, Many Others: Comparing Caregiver Attendance and Missed Treatment Hours in Pediatric Physical Therapy for Children With Cerebral Palsy. Phys Ther. 2025 Nov 29;105(12):pzaf131. doi: 10.1093/ptj/pzaf131. PMID 41206728
- [Derived] Scott KS, Barbosa GO, Pan J, Heathcock JC. Using the PODCI to Measure Motor Function and Parent Expectations in Children With Cerebral Palsy. Phys Ther. 2021 Dec 1;101(12):pzab215. doi: 10.1093/ptj/pzab215. PMID 34529078